CLINICAL TRIAL: NCT02756910
Title: Perioperative Accuracy of the Raiing Wireless Axillary Thermometer
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Lijian Pei, Associate Professor, Peking Union Medical College Hospital
Other Study IDs: HS-1019
Record Dates: First submitted 2016-04-03; First posted 2016-04-29 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-02

CONDITIONS: Major Surgery Under General Anesthesia
Keywords: open abdominal surgery; anesthesia, general

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery Patients >1.5 Hrs: Use esophageal catheter for core temperature monitoring, Foley catheter for bladder temperature monitoring, and iThermonitor (WT701) for axillary temperature monitoring
  Interventions: Device: iThermonitor (WT701)

INTERVENTIONS:
Device: iThermonitor (WT701) — Continuously monitor the axillary temperature during surgery

SUMMARY:
A new wireless axillary thermometer from Raiing Medical uses a proprietary system, iThermonitor (WT701), to provide better estimates of core temperature than a conventional axillary probe. Improvement results in part because the axillary probe measures and records temperatures continuously every 4 seconds and includes software to compensate for ambient temperature and positional changes including arm abduction.

Whether the iThermonitor is sufficiently accurate for clinical use remains unknown. The investigators thus propose to evaluate the system in perioperative patients who often experience thermal perturbations over a range of several °C. Specifically, the investigators propose to determine the precision and accuracy of iThermonitor in surgical patients and during the initial hour of recovery. As in previous studies, the investigators will consider the thermometer sufficiently accurate for clinical use if most Raiing temperatures are within ±0.5°C of the reference temperature.

DETAILED DESCRIPTION:
Patient characteristics, including age, height, weight, sex, and ASA status, and details of the surgery, including procedure and postoperative diagnosis will be recorded. The investigator will record the time of anesthesia induction and emergence. At 10-minute intervals during surgery, the investigator will record inspired volatile anesthetic concentration, mean-arterial pressure, type of thermal management device(s), and urine output over the previous 10-minute interval.

After induction of general anesthesia (without restriction as to type), the anesthesiologist will insert a temperature sensor into the distal esophagus. The distance will be determined by maximal heart sounds (if a stethoscope is used), or the probe will be inserted 0.48.(sitting height) - 4.4 cm. If an esophageal probe cannot be used, a thermometer can be inserted to between 10 and 20 cm into the nasopharynx. The surgical team will position a Foley catheter with temperature sensor into the urinary bladder. Ambient temperature will be recorded from an electronic probe situated at the height of the patients, well away from any heat-producing equipment.

Axillary temperature will be recorded by iThermonitor, a Raiing Medical wireless module, paired to an iPhone. An adhesive patch provided by Raiing will be used to securely position the Railing probe in a shaved axilla before the anesthesia induction. Patients will be asked to adduct the ipsilateral arm for up to 5 minutes after the probe is inserted, or until the temperature displayed on the paired iPhone is stable. Thereafter, patients will be free to move their arms.Monitored arm position during surgery will be recorded (arm tightly tucked, arm loose at side, arm abducted).

Temperatures will be recorded at 10-minute intervals during surgery and during the initial postoperative hour. Just before anesthetic emergence, the esophageal or nasopharyngeal thermometer will be removed, but the Foley catheter retained. The axillary device will then be removed after an hour of recovery, and the study concluded. The Foley catheter can be removed or retained per clinical need.

ELIGIBILITY:
Inclusion Criteria:

* adults having an American Society of Anesthesiologists (ASA) physical status of 1-3
* must be scheduled for surgery of the abdomen or pelvis that is expected to last 1.5-4 hours
* require general endotracheal anesthesia and insertion of a Foley catheter

Exclusion Criteria:

* patients in whom neither esophageal nor nasopharyngeal temperature monitoring is practical
* patients in whom active intravenous infusion is required in both arms
* patients who are allergic to hydrogel

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lijian Pei, MD, Principal Investigator — Associate Prof. of Dept. of Anesthesiology, PUMCH; Yuguang Huang, MD, Study Chair — Chair of Dept. of Anesthesiology, PUMCH; Daniel I Sessler, MD, Study Director — Chair of Dept. of Outcomes Research, Anesthesiology Institute, Cleveland Clinic
Locations (1):
- Dept. of Anesthesiology, PUMCH, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sessler DI. Temperature monitoring and perioperative thermoregulation. Anesthesiology. 2008 Aug;109(2):318-38. doi: 10.1097/ALN.0b013e31817f6d76. PMID 18648241
- [Background] Sessler DI. Perioperative heat balance. Anesthesiology. 2000 Feb;92(2):578-96. doi: 10.1097/00000542-200002000-00042. PMID 10691247
- [Background] Sessler DI. Complications and treatment of mild hypothermia. Anesthesiology. 2001 Aug;95(2):531-43. doi: 10.1097/00000542-200108000-00040. No abstract available. PMID 11506130
- [Background] Schmied H, Kurz A, Sessler DI, Kozek S, Reiter A. Mild hypothermia increases blood loss and transfusion requirements during total hip arthroplasty. Lancet. 1996 Feb 3;347(8997):289-92. doi: 10.1016/s0140-6736(96)90466-3. PMID 8569362
- [Background] Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. Study of Wound Infection and Temperature Group. N Engl J Med. 1996 May 9;334(19):1209-15. doi: 10.1056/NEJM199605093341901. PMID 8606715
- [Background] Lenhardt R, Marker E, Goll V, Tschernich H, Kurz A, Sessler DI, Narzt E, Lackner F. Mild intraoperative hypothermia prolongs postanesthetic recovery. Anesthesiology. 1997 Dec;87(6):1318-23. doi: 10.1097/00000542-199712000-00009. PMID 9416715
- [Background] Simon HB. Hyperthermia. N Engl J Med. 1993 Aug 12;329(7):483-7. doi: 10.1056/NEJM199308123290708. No abstract available. PMID 8332154
- [Background] Sessler DI. Malignant hyperthermia. J Pediatr. 1986 Jul;109(1):9-14. doi: 10.1016/s0022-3476(86)80563-7. No abstract available. PMID 3522838
- [Background] Sessler DI. A proposal for new temperature monitoring and thermal management guidelines. Anesthesiology. 1998 Nov;89(5):1298-300. doi: 10.1097/00000542-199811000-00061. No abstract available. PMID 9822041
- [Background] Bissonnette B, Sessler DI, LaFlamme P. Intraoperative temperature monitoring sites in infants and children and the effect of inspired gas warming on esophageal temperature. Anesth Analg. 1989 Aug;69(2):192-6. PMID 2764288
- [Background] Cork RC, Vaughan RW, Humphrey LS. Precision and accuracy of intraoperative temperature monitoring. Anesth Analg. 1983 Feb;62(2):211-4. PMID 6829923
- [Background] Sessler DI. Temperature monitoring and management during neuraxial anesthesia. Anesth Analg. 1999 Feb;88(2):243-5. doi: 10.1097/00000539-199902000-00003. No abstract available. PMID 9972734
- [Background] Amoateng-Adjepong Y, Del Mundo J, Manthous CA. Accuracy of an infrared tympanic thermometer. Chest. 1999 Apr;115(4):1002-5. doi: 10.1378/chest.115.4.1002. PMID 10208200
- [Background] Suleman MI, Doufas AG, Akca O, Ducharme M, Sessler DI. Insufficiency in a new temporal-artery thermometer for adult and pediatric patients. Anesth Analg. 2002 Jul;95(1):67-71, table of contents. doi: 10.1097/00000539-200207000-00012. PMID 12088945
- [Background] Harioka T, Matsukawa T, Ozaki M, Nomura K, Sone T, Kakuyama M, Toda H. "Deep-forehead" temperature correlates well with blood temperature. Can J Anaesth. 2000 Oct;47(10):980-3. doi: 10.1007/BF03024869. PMID 11032273
- [Background] Imamura M, Matsukawa T, Ozaki M, Sessler DI, Nishiyama T, Kumazawa T. The accuracy and precision of four infrared aural canal thermometers during cardiac surgery. Acta Anaesthesiol Scand. 1998 Nov;42(10):1222-6. doi: 10.1111/j.1399-6576.1998.tb05281.x. PMID 9834809
- [Background] Giuliano KK, Scott SS, Elliot S, Giuliano AJ. Temperature measurement in critically ill orally intubated adults: a comparison of pulmonary artery core, tympanic, and oral methods. Crit Care Med. 1999 Oct;27(10):2188-93. doi: 10.1097/00003246-199910000-00020. PMID 10548205
- [Background] Moran JL, Peter JV, Solomon PJ, Grealy B, Smith T, Ashforth W, Wake M, Peake SL, Peisach AR. Tympanic temperature measurements: are they reliable in the critically ill? A clinical study of measures of agreement. Crit Care Med. 2007 Jan;35(1):155-64. doi: 10.1097/01.CCM.0000250318.31453.CB. PMID 17095941
- [Background] Nussmeier NA, Cheng W, Marino M, Spata T, Li S, Daniels G, Clark T, Vaughn WK. Temperature during cardiopulmonary bypass: the discrepancies between monitored sites. Anesth Analg. 2006 Dec;103(6):1373-9. doi: 10.1213/01.ane.0000242535.02571.fa. PMID 17122206
- [Background] Robinson J, Charlton J, Seal R, Spady D, Joffres MR. Oesophageal, rectal, axillary, tympanic and pulmonary artery temperatures during cardiac surgery. Can J Anaesth. 1998 Apr;45(4):317-23. doi: 10.1007/BF03012021. PMID 9597204
- [Background] Webb GE. Comparison of esophageal and tympanic temperature monitoring during cardiopulmonary bypass. Anesth Analg. 1973 Sep-Oct;52(5):729-33. No abstract available. PMID 4542341
- [Background] Patel N, Smith CE, Pinchak AC, Hagen JF. Comparison of esophageal, tympanic, and forehead skin temperatures in adult patients. J Clin Anesth. 1996 Sep;8(6):462-8. doi: 10.1016/0952-8180(96)00103-1. PMID 8998260
- [Background] Lefrant JY, Muller L, de La Coussaye JE, Benbabaali M, Lebris C, Zeitoun N, Mari C, Saissi G, Ripart J, Eledjam JJ. Temperature measurement in intensive care patients: comparison of urinary bladder, oesophageal, rectal, axillary, and inguinal methods versus pulmonary artery core method. Intensive Care Med. 2003 Mar;29(3):414-8. doi: 10.1007/s00134-002-1619-5. Epub 2003 Feb 8. PMID 12577157
- [Background] Kaufman RD. Relationship between esophageal temperature gradient and heart and lung sounds heard by esophageal stethoscope. Anesth Analg. 1987 Oct;66(10):1046-8. No abstract available. PMID 3631570
- [Background] Mekjavic IB, Rempel ME. Determination of esophageal probe insertion length based on standing and sitting height. J Appl Physiol (1985). 1990 Jul;69(1):376-9. doi: 10.1152/jappl.1990.69.1.376. PMID 2394660
- [Background] Horrow JC, Rosenberg H. Does urinary catheter temperature reflect core temperature during cardiac surgery? Anesthesiology. 1988 Dec;69(6):986-9. doi: 10.1097/00000542-198812000-00037. No abstract available. PMID 3195774
- [Background] Tandberg D, Sklar D. Effect of tachypnea on the estimation of body temperature by an oral thermometer. N Engl J Med. 1983 Apr 21;308(16):945-6. doi: 10.1056/NEJM198304213081607. No abstract available. PMID 6835296
- [Background] Arkilic CF, Akca O, Taguchi A, Sessler DI, Kurz A. Temperature monitoring and management during neuraxial anesthesia: an observational study. Anesth Analg. 2000 Sep;91(3):662-6. doi: 10.1097/00000539-200009000-00031. PMID 10960396
- [Background] Langham GE, Maheshwari A, Contrera K, You J, Mascha E, Sessler DI. Noninvasive temperature monitoring in postanesthesia care units. Anesthesiology. 2009 Jul;111(1):90-6. doi: 10.1097/ALN.0b013e3181a864ca. PMID 19512860
- [Background] Giuliano KK, Giuliano AJ, Scott SS, MacLachlan E, Pysznik E, Elliot S, Woytowicz D. Temperature measurement in critically ill adults: a comparison of tympanic and oral methods. Am J Crit Care. 2000 Jul;9(4):254-61. PMID 10888148
- [Background] Insler SR, Sessler DI. Perioperative thermoregulation and temperature monitoring. Anesthesiol Clin. 2006 Dec;24(4):823-37. doi: 10.1016/j.atc.2006.09.001. PMID 17342966
- [Background] Erickson RS. The continuing question of how best to measure body temperature. Crit Care Med. 1999 Oct;27(10):2307-10. doi: 10.1097/00003246-199910000-00051. No abstract available. PMID 10548236
- [Background] Matsukawa T, Ozaki M, Hanagata K, Iwashita H, Miyaji T, Kumazawa T. A comparison of four infrared tympanic thermometers with tympanic membrane temperatures measured by thermocouples. Can J Anaesth. 1996 Dec;43(12):1224-8. doi: 10.1007/BF03013429. PMID 8955971
- [Background] Yaron M, Lowenstein SR, Koziol-McLain J. Measuring the accuracy of the infrared tympanic thermometer: correlation does not signify agreement. J Emerg Med. 1995 Sep-Oct;13(5):617-21. doi: 10.1016/0736-4679(95)00065-i. PMID 8530778
- [Background] Matsukawa T, Kashimoto S, Miyaji T, Hanagata K, Iriki M, Kumazawa T. A new infrared tympanic thermometer in surgery and anesthesia. J Anesth. 1993 Jan;7(1):33-9. doi: 10.1007/s0054030070033. PMID 15278493
- [Background] Greenes DS, Fleisher GR. Accuracy of a noninvasive temporal artery thermometer for use in infants. Arch Pediatr Adolesc Med. 2001 Mar;155(3):376-81. doi: 10.1001/archpedi.155.3.376. PMID 11231805
- [Background] Ikeda T, Sessler DI, Marder D, Xiong J. Influence of thermoregulatory vasomotion and ambient temperature variation on the accuracy of core-temperature estimates by cutaneous liquid-crystal thermometers. Anesthesiology. 1997 Mar;86(3):603-12. doi: 10.1097/00000542-199703000-00012. PMID 9066326
- [Background] Giuffre M, Heidenreich T, Carney-Gersten P, Dorsch JA, Heidenreich E. The relationship between axillary and core body temperature measurements. Appl Nurs Res. 1990 May;3(2):52-5. doi: 10.1016/s0897-1897(05)80158-2. PMID 2357072
- [Background] Lodha R, Mukerji N, Sinha N, Pandey RM, Jain Y. Is axillary temperature an appropriate surrogate for core temperature? Indian J Pediatr. 2000 Aug;67(8):571-4. doi: 10.1007/BF02758482. PMID 10984997
- [Background] Muma BK, Treloar DJ, Wurmlinger K, Peterson E, Vitae A. Comparison of rectal, axillary, and tympanic membrane temperatures in infants and young children. Ann Emerg Med. 1991 Jan;20(1):41-4. doi: 10.1016/s0196-0644(05)81116-3. PMID 1984726
- [Background] Ogren JM. The inaccuracy of axillary temperatures measured with an electronic thermometer. Am J Dis Child. 1990 Jan;144(1):109-11. doi: 10.1001/archpedi.1990.02150250121048. PMID 2294708
- [Background] Sund-Levander M, Forsberg C, Wahren LK. Normal oral, rectal, tympanic and axillary body temperature in adult men and women: a systematic literature review. Scand J Caring Sci. 2002 Jun;16(2):122-8. doi: 10.1046/j.1471-6712.2002.00069.x. PMID 12000664
- [Background] Matsukawa T, Sessler DI, Ozaki M, Hanagata K, Iwashita H, Kumazawa T. Comparison of distal oesophageal temperature with "deep" and tracheal temperatures. Can J Anaesth. 1997 Apr;44(4):433-8. doi: 10.1007/BF03014466. PMID 9104528
- [Background] Matsukawa T, Ozaki M, Sessler DI, Nishiyama T, Imamura M, Kumazawa T. Accuracy and precision of "deep sternal" and tracheal temperatures at high- and low-fresh-gas flows. Br J Anaesth. 1998 Aug;81(2):171-5. doi: 10.1093/bja/81.2.171. PMID 9813517
- [Background] Eshraghi Y, Nasr V, Parra-Sanchez I, Van Duren A, Botham M, Santoscoy T, Sessler DI. An evaluation of a zero-heat-flux cutaneous thermometer in cardiac surgical patients. Anesth Analg. 2014 Sep;119(3):543-549. doi: 10.1213/ANE.0000000000000319. PMID 25045862
- [Background] Sessler DI, Lee KA, McGuire J. Isoflurane anesthesia and circadian temperature cycles in humans. Anesthesiology. 1991 Dec;75(6):985-9. doi: 10.1097/00000542-199112000-00010. PMID 1741520
- [Background] Winkler M, Akca O, Birkenberg B, Hetz H, Scheck T, Arkilic CF, Kabon B, Marker E, Grubl A, Czepan R, Greher M, Goll V, Gottsauner-Wolf F, Kurz A, Sessler DI. Aggressive warming reduces blood loss during hip arthroplasty. Anesth Analg. 2000 Oct;91(4):978-84. doi: 10.1097/00000539-200010000-00039. PMID 11004060

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgery Patients >1.5 Hrs
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Surgery Patients >1.5 Hrs
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 45

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of iThermonitor in Surgical Patients
Description: Accuracy, defined as the true difference between reference and iThermonitor temperature. The esophageal temperature will be the core temperature reference during surgery.
  The primary outcome measure is the proportion of iThermonitor measurements for a patient that are within 0.5° C of the reference will be calculated, and this proportion (median, quartiles, 95% CI) will be summarized across patients.
  The Secondary outcome measure are bias and 95% CIs determined by repeated-measures Bland-Altman analysis.
  For each patient the average difference between the iThermometer and the reference temperature will be calculated. Patient iThermonitor measurements will be regressed on patient reference measurements to assess the Pearson correlation and 95% CI between iThermonitor and reference and to estimate the bias (slope) of device versus reference.
Time Frame: From 1 to 3 hours after induction of anesthesia
Population: There were a total of 3,339 sets of iThermonitor and reference measurements from 80 patients (42 sets per patient on average). The iThermonitor temperature and the reference esophageal temperature agreed well overall. The iThermonitor temperatures ranged from 34.7 to 38.3°C, while the esophageal core temperatures ranged from 34.6 to 37.9°C
Measure: Mean (Standard Deviation); unit: celsius
Arm/Group | Surgery Patients >1.5 Hrs
Number analyzed (Participants) | 80
celsius | 0.14 (0.26)
Statistical Analysis 1: Comparison: Surgery Patients >1.5 Hrs; Test type: Other; p < 0.05, bootstrapping; percentile method = 0.5, Standard Deviation 1.96

ADVERSE EVENTS:
Time Frame: During the operation
Description: Skin and Subcutaneous Tissue Disorders：skin crush
Arm/Group | Surgery Patients >1.5 Hrs
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No